CLINICAL TRIAL: NCT03356847
Title: Evaluation of the Rotational Stability of the Monofocal SISA Implant Following Cataract Surgery
Acronym: SISALens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDIL/2017/DM-01
Record Dates: First submitted 2017-09-29; First posted 2017-11-29 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2017-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SISA implant (Experimental)
  Interventions: Device: Fitting of ocular implant

INTERVENTIONS:
Device: Fitting of ocular implant — Removal of natural lens and replacement with a SISA monofocal intraocular implant

SUMMARY:
A good efficacy as well as good rotary stability is expected with the ocular implant.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient must be available for 6 months follow-up
* The patient it aged at least 18 years
* Patient requires surgery for cataracts with removal of the opacified natural lens and replacement with the SISA implant, according to standard procedure
* The surgery is elective
* The patient has clear and non-pathological corneas
* The patient needs an implant strength (LIO) between +10D and +30D
* Corneal astigmatism less than or equal to 1.50D in the eye to be operated (or cataract eye

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice or state guardianship
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is pregnant or breastfeeding
* The patient has other ocular comorbidities with poor visual acuity prognosis postoperatively
* Previous ocular trauma or surgery
* Dilation of the pupil <7mm with mydriatic drugs
* Implantation with a rhexis that does not cover the optic of the implant by more than 1 cadranel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Rotational stability of SISA monofocal implant following cataracts surgery | 4 Months
  rotation in degrees measured by Labview software

SECONDARY OUTCOMES:
Rotational stability of SISA monofocal implant following cataracts surgery | Day 0
  rotation in degrees measured by Labview software
Rotational stability of SISA monofocal implant following cataracts surgery | Day 7
  rotation in degrees measured by Labview software
Rotational stability of SISA monofocal implant following cataracts surgery | 1 Month
  rotation in degrees measured by Labview software
Centering of SISA monofocal implant | Day 0
  Distance in mm between centers of the coreal and optic ellipses
Centering of SISA monofocal implant | Day 7
  Distance in mm between centers of the coreal and optic ellipses
Centering of SISA monofocal implant | Month 1
  Distance in mm between centers of the coreal and optic ellipses
Centering of SISA monofocal implant | Month 4
  Distance in mm between centers of the coreal and optic ellipses
Refractive precision | Day 7
  Early Treatment Diabetic Retinopathy Study scale; chart 1 at 4 meters; diopters
Refractive precision | Month 1
  Early Treatment Diabetic Retinopathy Study scale; chart 1 at 4 meters; diopters;
Refractive precision | Month 4
  Early Treatment Diabetic Retinopathy Study scale; chart 1 at 4 meters; diopters
Visual acuity with and without correction | Day 7
  Early Treatment Diabetic Retinopathy Study scale, logMAR
Visual acuity with and without correction | Month 1
  Early Treatment Diabetic Retinopathy Study scale, logMAR
Visual acuity with and without correction | Month 4
  Early Treatment Diabetic Retinopathy Study scale, logMAR
Perioperative complications | Day 0
  Yes/no
Postoperative complications | Day 7
  Yes/no
Occurrence of undesirable events, | Day 0
  Presence/absence of each event, including, but not limited to: inflammation, retinal detachment, macular edema, corneal endothelial lesion,corneal edema, implant gets decentred or tilted,
Occurrence of undesirable events, | Day 7
  Presence/absence of each event, including, but not limited to: inflammation, retinal detachment, macular edema, corneal endothelial lesion,corneal edema, implant gets decentred or tilted,
Occurrence of undesirable events, | Month 1
  Presence/absence of each event, including, but not limited to: inflammation, retinal detachment, macular edema, corneal endothelial lesion,corneal edema, implant gets decentred or tilted,
Occurrence of undesirable events, | Month 7
  Presence/absence of each event, including, but not limited to: inflammation, retinal detachment, macular edema, corneal endothelial lesion,corneal edema, implant gets decentred or tilted,

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France